CLINICAL TRIAL: NCT03396536
Title: The Impact of Peri-implant Soft Tissue Properties on Patient-reported and Clinically Assessed Outcomes: A Prospective Study
Brief Title: The Impact of Peri-implant Soft Tissue Properties on Patient-reported and Clinically Assessed Outcomes
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Other Study IDs: 11003
Record Dates: First submitted 2017-12-08; First posted 2018-01-11 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Keratinized Mucosa
Keywords: implant; oral hygiene; discomfort

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group 1 will be implants with keratinized mucosa (KM).
  Interventions: Other: Evaluation of KM
- Group 2: Group 2 implants without keratinized mucosa (KM). Alveolar mucosa (AM) directly present around the implant.
  Interventions: Other: Evaluation of KM

INTERVENTIONS:
Other: Evaluation of KM — KM will be evaluated. The alveolar mucosa will be stained with Lugol's solution, by means of a cotton swab. A cotton roll will be soaked in the solution and gently applied on the mucosa around the implant. Since Lugol's solution is selective to the glycogen present in AM, the muco-gingival junction as the borderline between the blue-stained alveolar mucosa and KM can be easily identified.
  A manual periodontal probe with 1 mm markings will measure the distance from the peri-implant margin and the muco-gingival junction.
  Mucosal thickness (MT) will be measured after topical application of the anesthetics. MT will be evaluated inserting a 27G needle with a rubber stop 1 mm below the peri-implant mucosal margin at the mid-buccal aspect, until the abutment is engaged. The needle will be removed and the distance between the rubber stop and the point of the needle will be measured with a manual periodontal probe.

SUMMARY:
The objective of this study is to evaluate patient discomfort while performing oral hygiene (OH) around implants with and without keratinized mucosa (KM) and assess peri-implant soft tissue esthetic satisfaction and other clinical parameters at the 3- and 6-month follow-up visits. Group 1 will be implants with KM and Group 2 implants without KM. The hypotheses underlying this proposal are (1) that dental implants surrounded by KM will have better patient-reported outcomes regarding discomfort during brushing compared with those that lack KM; (2) that dental implants with KM will show more favorable clinical outcomes (plaque index, bleeding on probing, pocket depth and peri-implant recession) compared with those without KM and (3) that dental implants with KM will have higher patient peri-implant tissue esthetic satisfaction compared with those without KM.

DETAILED DESCRIPTION:
In the oral cavity, the soft tissue of the alveolar ridge can be classified as keratinized mucosa (KM) or alveolar mucosa (AM). Typically KM forms a cuff around an implant, while AM is farther away and covers the alveolar ridge, as well the lips, the inside of the cheeks, the floor of the mouth under the tongue. KM is pink in color and has a keratinized epithelium. AM is red and has a non-keratinized epithelium. Due to anatomical or surgical reasons KM on the buccal site might be missing. Therefore implants without KM have AM directly around their collar. The two groups in the research will be defined according to the presence or absence of KM. Group 1 will be implants with KM and Group 2 implants without KM. In Group 2 AM will be directly present around the implant.

Although specific situations recommend a minimal width of 2 mm of keratinized tissue around teeth to prevent gingival inflammation, the influence of keratinized tissue on peri-implant clinical and patient-reported outcomes still needs to be investigated. Many authors have stated that that the presence of peri-implant keratinized mucosa is a prerequisite for the maintenance of soft tissue health and have advocated for soft tissue augmentation procedures around implants. Nevertheless, since other authors failed to demonstrate a significant association between clinical inflammatory parameters and the quality of peri-implant mucosa, soft tissue augmentation procedures are not recommended, unless the patient reports pain and discomfort while brushing around an implant without KM or unless there are esthetic concerns. Those recommendations are however not evidence-based. To the best of our knowledge no prospective studies have been conducted to evaluate systematically discomfort during brushing at implant sites and patient soft tissue esthetic assessment, with special emphasis on the quality of peri-implant soft tissue.

Dental implants can be placed according to a one-stage or a two-stage protocol. For two-stage implant surgery, as is required for this study, there are the following steps (stages).

1. Implant placement surgery occurs. At this time, the implant is placed in the bone. A cover screw is placed on top of the implant and then covered with mucosa (gums).
2. After a period of a few months to allow for healing, the mucosa (gums) on top of the implant is opened making a small incision. The cover screw is removed. Then, an additional implant piece called a healing abutment is placed that penetrates through the gums. This healing abutment allows for soft tissues to heal around the implant abutment before an impression is made for the manufacture of the implant crown.

Additional steps are then required for placement of the implant crown (artificial tooth). For this study, the baseline visit will be at the time of step 2. The implant will already have been placed previously and the patient will be returning to the clinic for their scheduled second stage surgery.

Discomfort while brushing at an implant site is a parameter that clinical trials should include. In a recent study it was reported that 6 patients out of 16 reported discomfort while brushing implants without KM, while no patients reported discomfort while brushing in the group of implants with KM. Higher plaque accumulation was also found around implants without KM. In this study, however, there were some limitations, such as a lack of standardization in terms of OH instructions and absence of adequate description of the outcome discomfort. Finally an esthetic evaluation of the implant-supported restoration was not reported. Since patient esthetic evaluation on the appearance of the soft tissue is less optimal than the overall esthetic evaluation and esthetic concerns might justify soft tissue augmentation procedures around implants, further prospective studies should be focused on patient soft tissue esthetic assessment.

A survey was conducted to assess the validity and the reliability of a visual analogue scale (VAS) for discomfort during brushing at implant site and VAS for esthetic satisfaction of the soft tissue around implants (IRB #10863 Testing the validity and reliability of a survey to record discomfort during brushing around dental implants and patient-assessed soft tissue esthetic satisfaction at implant-supported restorations). The face and content validity of the scales was assessed by showing them to 5 lay people and 5 postgraduate residents in the Department of Periodontology at Tufts University School of Dental Medicine. The five lay people were asked whether the questions on both surveys were phrased appropriately, and whether the scales were clear. All subjects answered positively. The 5 postgraduate residents reported that VAS was the appropriate method to measure the variable "discomfort while brushing around implants" and to measure patient-assessed soft tissue esthetic satisfaction. However, for both the 10 cm VAS scales, the majority of subjects (lay people and residents) pointed out that there was a lack of directionality. Therefore it was decided to add numbers to the scales. For discomfort during brushing the scale had on the left side displayed as 0 the absence of discomfort and on the right as 10 the maximum discomfort. For esthetic satisfaction, the left side of the scale represented no satisfaction as 0, while 10 at the right end of the scale represented extreme satisfaction.

Fifteen (15) patients in the Department of Periodontology at Tufts University School of Dental Medicine were recruited to assess the reliability of the VAS scales for discomfort during brushing and for soft tissue esthetic satisfaction at implant sites. The following question was asked: "If the left side of the scale is the absence of discomfort and the right side of the scale is extreme discomfort, how much discomfort do you have while brushing around your implant?". The question for the second VAS was: "If the left side of the scale is no satisfaction and the right side of the scale is extreme satisfaction, how satisfied are you with the appearance of the gums around your implant?". The patient marked a line with a fine point marker or pen at the level of one of the numbers below the scales. The reliability of the instruments was tested using the test-retest method, administrating the survey instruments to the same subjects at a time difference of 30 minutes. Fourteen and 12 subjects had the same results on both the first and second survey for discomfort during brushing and soft tissue esthetic satisfaction. Therefore the 2 scales were considered a reliable method to record the outcome of interests.

The main objective of this study is to define, for the first time, whether the presence of KM around dental implants is required from both patients' and clinicians' perspectives, a concept with important clinical implications that has been the source of controversy in the field. The need to include patient-reported outcomes (PROs) in implant dentistry has been emphasized in many recently published reviews. Because patients ultimately seek professional care to improve their own quality of life, optimal care is achieved not only if some specific clinical standards are met, but also if patient expectations are satisfied and their quality of life is improved. Indeed, in an evidence-based approach, it is important to address these aspects of treatment as well. The impact of this study will be high, since its successful execution will provide a rationale for using soft tissue augmentation procedures in implant therapy, based on PROs and other clinical assessed outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients treatment planned for second stage implant surgery (having already had stage one completed
* Partially or fully edentulous patients that have a single implant or have multiple implants that are non-adjacent
* Patients that have implant(s) that will be restored with fixed cement- or screw-retained restoration(s)

Exclusion Criteria:

* Unwilling to sign informed consent form
* Non-English speaking subjects
* Pregnant women (self-reported)
* Heavy smokers (10 cigarettes/day)
* Known allergy to iodine and/or potassium iodide (ingredients of Lugol's solution)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A sample size calculation was conducted using nQuery Advisor (Version 7.0). Assuming that 37.5% in the non-KM group (Group 2) have high discomfort and 2% in the KM Group (Group 1) have high discomfort, a Type I error rate of 5%/2 = 2.5% per test and a power of 80% are obtained as long as there are n=23 subjects with a KM implant and n=23 subjects with a non-KM implant. To account for possible dropout, up to n=28 subjects with each type of peri-implant mucosa group (for a total of up to 56 subjects) will be included in the study. Up to 80 subjects will be enrolled in order to have 56 complete the study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2015-06-09 (Actual); Study Completion 2015-06-09 (Actual)

PRIMARY OUTCOMES:
Patient Discomfort | Change in patient discomfort at 3 months
  This will be a prospective clinical study to evaluate patient discomfort while performing oral hygiene (OH) around implants with and without KM and assess peri-implant soft tissue esthetic evaluation and other clinical parameters at the 3- and 6-month follow-up visits. The primary outcome will be discomfort during brushing at implant site.
Patient Discomfort | Change in patient discomfort at 6 months
  This will be a prospective clinical study to evaluate patient discomfort while performing oral hygiene (OH) around implants with and without KM and assess peri-implant soft tissue esthetic evaluation and other clinical parameters at the 3- and 6-month follow-up visits. The primary outcome will be discomfort during brushing at implant site.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Weber, Principal Investigator — TUSDM

IPD SHARING:
Plan to Share IPD: No